CLINICAL TRIAL: NCT06935474
Title: Multi-center, Phase 1/2 Study of an Autologous Anti-CD20/BCMA CAR T Cell Therapy (C-CAR168) for the Treatment of Autoimmune Disease Refractory to Standard Therapy
Brief Title: C-CAR168 CAR T Cell Therapy for Refractory Autoimmune Disease
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbelZeta Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABZT-411
Record Dates: First submitted 2025-03-26; First posted 2025-04-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Lupus Nephritis (LN)
Keywords: Autoimmune; Lupus Nepritis; Systemic Lupus Erythematosus; CAR-T; CD20; C-CAR168; BCMA
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: This study uses a 3+3 dose escalation design to determine the Maximum Tolerated Dose (MTD) and/or Recommended Dose (RD) of C-CAR168. Subjects in each dose level will be enrolled sequentially with a minimum 28-day interval between infusions. Upon completion of dose escalation, 12-24 additional subjects may be enrolled in a dose expansion phase, pending Safety Review Committee (SRC) approval. No staggering is required during the expansion phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 2: Dose Level 1 (DL1) (Experimental): Dose: 0.75 × 10⁶ CAR+ cells/kg Starting dose for escalation phase. First 3 subjects must be staggered by 28 days.
  Interventions: Biological: C-CAR168
- Arm 3: Dose Level 2 (DL2) (Experimental): Dose: 1.5 × 10⁶ CAR+ cells/kg Second dose level in escalation phase. Subject enrollment staggered by 28 days.
  Interventions: Biological: C-CAR168
- Arm 1: Dose Level -1 (DL-1) (Experimental): 0.5 × 10⁶ CAR+ cells/kg Optional dose level, administered only upon Safety Review Committee (SRC) recommendation.
  Interventions: Biological: C-CAR168
- Arm 4: Dose Level 3 (DL3) (Experimental): Dose: 2.0 × 10⁶ CAR+ cells/kg Optional dose level pending SRC review and approval.
  Interventions: Biological: C-CAR168
- Arm 5: Dose Expansion Cohort (Experimental): Dose: To be selected based on MTD/RD identified in escalation phase. 12-24 additional subjects will be treated at the selected dose level. No staggered dosing required.
  Interventions: Biological: C-CAR168

INTERVENTIONS:
Biological: C-CAR168 — This is a multi-center, Phase 1/2, open-label, dose-escalation and dose-expansion study evaluating C-CAR168 for the treatment of autoimmune diseases refractory to standard therapy. A traditional 3+3 design is used to identify the Maximum Tolerated Dose (MTD) and/or Recommended Dose (RD) in disease-specific cohorts.

SUMMARY:
This multi-center, open-label, Phase 1/2 study aims to evaluate the safety, tolerability, and preliminary efficacy of C-CAR168, an autologous anti-CD20/BCMA CAR-T therapy, in patients with autoimmune diseases refractory to standard treatments. The study includes both dose escalation and dose expansion phases, with participants grouped into condition-specific cohorts.

The purpose of this study is to:

1. Test the safety and ability for subjects with autoimmune refractory to standard treatment to tolerate the C-CAR168.
2. Determine the recommended Phase 2 dose of C-CAR168 in subjects with autoimmune disease refractory to standard treatment.

Participants will be asked to:

* Undergo screening to determine eligibility based on entry criteria.
* Taper steroid use before leukapheresis.
* Undergo leukapheresis for the manufacturing of C-CAR168.
* Temporarily discontinue immunosuppressive therapy at least 7 days prior to leukapheresis.
* Receive bridging therapy (steroids) if necessary to maintain disease stability during C-CAR168 manufacturing.
* Undergo lymphodepletion therapy with fludarabine and cyclophosphamide.
* Receive a single intravenous infusion of C-CAR168 at the assigned dose level on Day 0.
* Attend regular safety and efficacy assessments for up to 24 months post-infusion.
* Undergo dose-limiting toxicity evaluation during the first 28 days post-infusion (for those in the dose escalation phase).
* Follow withdrawal procedures if necessary, including a discharge visit within 14 days if their condition deteriorates, unacceptable toxicity occurs, they no longer meet criteria, or they choose to withdraw.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent: Voluntary signed consent required.
2. Age & Gender: Males and females, 18-70 years old.
3. Diagnosis: Clinical diagnosis of SLE per EULAR/ACR criteria for at least 6 months.
4. Lupus Nephritis (LN): Biopsy-confirmed active proliferative LN (Class III/IV ± V) within the past 12 months.
5. Refractory Disease:

   * Treated with at least two immunosuppressants for ≥8 weeks.
   * Stable but active disease despite standard therapy (steroids, IS, monoclonal antibodies).
   * Steroid dose ≤30 mg/day (if applicable).
6. Disease Activity at Screening:

   * SLE without LN: SLEDAI-2K ≥8 and 1 BILAG A or 2 BILAG B scores.
   * LN Patients: Proteinuria ≥1.0 g/day or UPCR ≥1.0 g/g.
7. Autoantibody Status:

   o Positive ANA (≥1:80), anti-dsDNA (≥30 IU/mL), and/or anti-Smith antibody.
8. Infection Status: No active infection within 2 weeks before leukapheresis.
9. Life Expectancy: Greater than 6 months.
10. Adequate Organ Function:

    * Bone Marrow: ANC ≥1.0×10⁹/L, ALC ≥0.5×10⁹/L, Hb ≥80 g/L, PLT ≥75×10⁹/L.
    * Coagulation: INR/APTT ≤1.5×ULN.
    * Cardiac: LVEF ≥45% by ECHO/MUGA.
    * Pulmonary: SpO₂ ≥92% on room air.
    * Liver: ALT/AST ≤2.5×ULN, total bilirubin <2.0 mg/dL.
    * Renal: Creatinine clearance ≥40 mL/min (Cockcroft-Gault).
11. Pregnancy & Contraception:

    * Women of childbearing potential must have a negative pregnancy test at screening.
    * Both male and female participants must use highly effective contraception for 1 year post-treatment.

Exclusion Criteria:

1. Any other concomitant diseases requiring long term systemic steroids (oral or intravenously) treatment that may confound the interpretation of study results or have interference with background steroid tapering for the subjects.
2. Any of the following:

   * Positive for Hepatitis B surface antigen (HBsAg)/core antibody (HBcAb)/e antibody (HBeAb)/e antigen (HBeAg).
   * Positive for Hepatitis C Virus (HCV) antibodies.
   * Positive for Human Immunodeficiency Virus (HIV) antibodies.
   * Positive for syphilis antigen or antibody.
3. Have an uncontrolled active infection.
4. History of major organ transplantation (such as heart, lung, liver, kidney) or history of bone marrow/hematopoietic stem cell transplantation.
5. History of any of stroke, unstable angina, myocardial infarction, congestive heart failure (NYHA Class III or IV), severe cardiomyopathy or ventricular arrhythmia requiring medication or mechanical control within 6 months of screening.
6. History of ≥ Grade 2 bleeding within the past 30 days.
7. Received a live vaccine within 4 weeks prior to signing the ICF.
8. Received any of the following treatments:

   * Prednisone treatment of ≥ 100 mg/d or equivalent corticosteroid therapy for ≥14 days within the previous 8 weeks.
   * Receive plasma exchange, plasma separation, hemodialysis, or intravenous injection of immunoglobulin (IVIG) within 14 days prior to leukapheresis.
   * Use of any other investigational clinical study drug within 28 days prior to leukapheresis. However, if the subject is not responsive to the treatment or have progressed and at least 3 half-lives have passed before the leukapheresis, he/she could be enrolled.
   * Previously received any CAR-T cell products or other genetically modified T cell therapies.
   * Rituximab/ocrelizumab/obinutuzumab within 6 months prior to screening
9. Pregnant or breastfeeding women.
10. History of seizure disorder, cerebrovascular ischemia/hemorrhage, dementia or cerebellar disease or other severe neuropsychiatric syndromes.
11. History of deep vein thrombosis or pulmonary embolism within six months of infusion (line associated DVT is allowed)
12. Diagnosed with malignant tumors within 5 years prior to signing the ICF, with the following exceptions: non-melanoma skin cancer that has been treated with radical therapy, localized prostate cancer, biopsy-confirmed cervical carcinoma in situ or squamous intraepithelial lesions detected by cervical smear, and completely excised breast carcinoma in situ.
13. Poor compliance, unwilling or unable to adhere to the study protocol based on the investigator's assessment.
14. Allergies to fludarabine, cyclophosphamide and/or known allergies to excipients of C-CAR168 cell product.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events or Dose Limiting Toxicities | Up to 24 months
  The number and severity of Adverse Events (AE) and Serious Adverse Events (SAE), including dose limiting toxicities (DLTs) will be recorded.

SECONDARY OUTCOMES:
To evaluate the efficacy of C-CAR168 | Up to 24 months
  Proportion of subjects meeting the KDIGO 2024 Clinical Practice Guidelines' Definition of Remission, which includes complete response, primary efficacy renal response, or partial response.
To evaluate the efficacy of C-CAR168 | Up to 24 months
  Proportion of subjects achieving SLEDAI-2K response over time.
To evaluate the efficacy of C-CAR168 | Up to 24 months
  Proportion of subjects achieving British Isles Lupus Assessment Group (BILAG)(BILAG) response over time.
Renal Related Events | Up to 24 months
  Record any renal related events during the study, including disease flare and the time to the event.
Time to Response | Up to 24 months
  The number of days to response from the infusion of C-CAR0168 to the first recorded remission.
Corticosteroid use | Up to 24 months
  The number of patients who achieved a low dose of steroids or no longer require.
To characterize the cellular kinetics of C-CAR168 | Up to 24 months
  Level of C-CAR168 positive cells in the blood.
To assess immunogenicity of C-CAR168 | Up to 24 months
  Presence of C-CAR168 antibodies.
To evaluate the efficacy of C-CAR168 | Up to 24 months
  Proportion of subjects whose for Physician Global Assessment (PGA) score does not worsen over time.
To evaluate the efficacy of C-CAR168 | Up to 24 months
  Proportion of subjects achieving a predefined score on the Visual Analog Scale (VAS) at specified time points.
  Efficacy will be assessed by evaluating changes in pain intensity as perceived by subjects, using the Visual Analog Scale (VAS). Subjects will rate their pain intensity on a scale from 0 (no pain) to 10 (worst imaginable pain). This will provide a subjective measure of pain severity over the course of the study.
To assess changes for reported health-related quality of life, overall health status | Up to 24 months
  To assess changes from baseline for Functional Assessment of Chronic Illness Therapy (FACIT).
  The 13-item questionnaire will measure the level of fatigue and its impact on daily functioning. Higher scores reflect less fatigue and better overall energy levels.
To assess changes for reported health-related quality of life, overall health status | Up to 24 months
  To assess changes from baseline for SF-36 (Short Form Health Survey). Efficacy will be assessed by evaluating changes in quality of life using the SF-36. Higher scores indicate better overall health and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Antonia, Principal Investigator — Duke University
Locations (1):
- AbelZeta, Inc., Rockville, Maryland, United States